CLINICAL TRIAL: NCT00969826
Title: A Clinical Study to Investigate the Pharmacokinetics and Pharmacodynamics of GCPGC After Single Subcutaneous Administration in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of a Novel Pegylated Recombinant Human Granulocyte-Colony Stimulating Factor
Acronym: GCPGC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Young-Joo Ahn, Clinical Research Team / Development Division Associate Director
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUCPT08_GCPGC
Record Dates: First submitted 2009-08-29; First posted 2009-09-01 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: GCPGC; Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GCPGC 30 μg/kg (Experimental): Ten volunteers were administered GCPGC 30 μg/kg or placebo (active:placebo=8:2)
  Interventions: Drug: GCPGC, Neulasta, Placebo
- GCPGC 100 μg/kg (Experimental): Ten volunteers were administered GCPGC 100 μg/kg or placebo (active:placebo=8:2)
  Interventions: Drug: GCPGC, Neulasta, Placebo
- GCPGC 300 μg/kg (Experimental): Ten volunteers would be administered GCPGC 300 μg/kg or placebo (active:placebo=8:2)
  Interventions: Drug: GCPGC, Neulasta, Placebo
- Neulasta 100 μg/kg (Experimental): Eight volunteers were administered Neulasta 100 μg/kg
  Interventions: Drug: GCPGC, Neulasta, Placebo

INTERVENTIONS:
Drug: GCPGC, Neulasta, Placebo — A single subcutaneous administration of GCPGC 30 μg/kg, GCPGC 100 μg/kg, GCPGC 300 μg/kg, placebo or Neulasta 100 μg/kg
  Other Names: Neulasta® (Amgen, USA; active comparator)

SUMMARY:
This study is a four arm, parallel study.

Ten were administered a single subcutaneous administration of 30, 100 and 300 μg/kg of GCPGC or placebo for each group (active:placebo=8:2). Eight were administered a single subcutaneous administration of 100 μg/kg of Neulasta (an active comparator).

DETAILED DESCRIPTION:
Eligibility for participation of this study was determined from demographic information, medical history, physical examination, electrocardiogram (ECG) and clinical laboratory tests within 3 weeks before study drug administration. Subjects suitable for this study were admitted to the Clinical Trials Center, Seoul National University Hospital on the day before dosing, and they were overnight-fasted from 10 p.m. of Day -1. Subjects were dosed study drug via subcutaneous around at 9 a.m. of Day 1. Subjects performed scheduled procedures including clinical laboratory tests, electrocardiograms and pharmacokinetic and pharmacodynamic samplings. Subjects were discharged on Day 8, and visited Clinical Trials Center on Day 9, Day 11 and Day 14. Study participation was terminated on post-study visit (Day 20 - 22).

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 20 to 40 years of age, inclusive (Age based on the date to give the informed consent)
* Weight: Between 60 - 75 kg, within ±20% of ideal body weight
* Normal clinical laboratory findings, especially for ANC value between 2000 to 7500, inclusive
* Subject who are reliable and willing to make themselves available during the study period, are willing to follow the study protocol, and give their written informed consent voluntarily

Exclusion Criteria:

* History of hypersensitive reaction to medication (aspirin, antibiotics)
* History of significant clinical illness needs medical caution, including cardiovascular, immunologic, hematologic, neuropsychiatric, respiratory, gastrointestinal, hepatic, or renal disease or other chronic disease
* History or evidence of drug abuse
* Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
* Participation in clinical trials of any drug within 60 days prior to the participation of the study
* Donation of whole blood within 60 days or a unit of blood within 30 days prior to the start of study
* Judged to be inappropriate for the study by the investigator

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Blood concentration of pegfilgrastim for pharmacokinetics | pre-dose, 3, 6, 9, 12, 24(2d), 36, 48(3d), 72(4d), 96(5d), 120(6d), 144(7d), 168(8d), 192h(9d), 240(11d), 312(14d)

SECONDARY OUTCOMES:
Absolute Neutrophil Count (ANC) | pre-dose, 6, 12, 24(2d), 48(3d), 72(4d), 96(5d), 120(6d), 144(7d), 168(8d), 192h(9d), 240(11d), 312(14d)
CD34+ Cell count | pre-dose, 6, 12, 24(2d), 48(3d), 72(4d), 96(5d), 120(6d), 144(7d), 168(8d), 192h(9d), 240(11d), 312(14d)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University College of Medicine and Hospital
Locations (1):
- Clinical Trials Center, Seoul National University Hospital, Seoul, South Korea